CLINICAL TRIAL: NCT03519035
Title: Study of Prevalence and Characteristics of Hallucinations in Patients With Borderline Personality Disorder
Brief Title: Study of Hallucinations in Patients With Borderline Personality Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0035; 2018-A00251-54 (Other: ID-RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Borderline Personality Disorder
Keywords: borderline; hallucinations; dissociation; post-traumatic stress disorder
MeSH Terms: conditions — Borderline Personality Disorder; Hallucinations; Dissociative Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Borderline personality disorder Patient: Patients will be recruited in the different services. They have to respect inclusion criteria which are : patient with BPD (clinical diagnosis), patients 18 years of age or older, patients who can give their consent.
  In this study, patients will have to pass different questionnaires (DIB-R, DES II, THQ, PCL-S, PSAS, qualitative questionnaire) in order to compare the characteristics between BDL patients with and without hallucinations.
  Interventions: Other: To pass different questionnaires

INTERVENTIONS:
Other: To pass different questionnaires — Patients will have to pass different questionnaires (DIB-R, DES II, THQ, PCL-S, PSAS, qualitative questionnaire) in order to compare the characteristics between BDL patients with and without hallucinations.

SUMMARY:
Hallucinations in borderline personality disorder are a frequent an serious trouble which have an important impact in patients lives. Despite this, they are often ignored by nursing staff, and are not an important criteria in Diagnostic and Statistical Manual (DSM) 5 and Classification Internationale des maladies (CIM-10). The main objective of our study is to assess the prevalence of this trouble in borderline personality disorder (BPD) population, and to characterize the hallucinations in order to compare our results with those of international studies.

DETAILED DESCRIPTION:
The borderline personality disorder (BPD) is a very common personality disorder which concerns about 1.35% of total population. It is characterized by an affective, emotional, social and professional instability and an important association with comorbidities like mood disorders, post-traumatic stress disorder, addictive problems and suicide mortality. Hallucinations seem to be frequent in this personality disorder, but are not often taken in consideration by nursing staff because of massive need of attention of this kind of patient. At this moment there is no study of prevalence of this trouble in France in free environment. In the same way, there is no qualitative study about hallucinations. That is why we can do a lot of progress in this part of psychiatry.

This research is an observational study of descriptive type. Patients will be recruited in the different services. In this study, patients will have to pass different questionnaires (DIB-R, DES II, THQ, PCL-S, PSAS, qualitative questionnaire) in order to compare the characteristics between BDL patients with and without hallucinations.

For that, the investigator will meet each patient twice, after information by the medical staff of the service and consent. During the first meeting, the investigator will get the socio-demographic characteristics, the verification of inclusion and non-inclusion criteria, and the DIB-R questionnaire to know if the patient has really BPD and hallucinations or not. This is the same interview for all patients. During the second meeting, we will look for dissociative symptoms with DES II questionnaire, then traumatic symptoms and post-traumatic stress disorder with THQ and PCL-S. The PSAS and qualitative questionnaire will be used for BPD patients with hallucinations.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and under 75
* Patient with borderline personality disorder (formerly or newly diagnosed diagnosis)
* Patient having given his opposition to his participation in research

Exclusion Criteria:

* Schizophrenia
* Major depressive episode characterized in progress
* Manic or hypomanic episode in progress
* History of head trauma
* Stroke, Parkinson's disease, dementia
* Autism
* Mental retardation
* Patient under the age of 75
* Patient who does not read or speak French
* Patient unable to give consent (includes protected persons: guardianship, trusteeship)
* Incarcerated patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with borderline personnality disorder (BPD) and they will be recruited in the different services.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of hallucination | 1 day
  During the first interview with the passage of the DIB-R scale It consists of determining whether or not hallucinations have occurred during the patient's life. This criterion will allow the outcome of the study to estimate the prevalence (over the last two years (as specified by the DIB-R questionnaire) but also over the lifetime to obtain additional data) hallucinatory manifestations in patients with a BDL course.
  All patients will have the same first interview, with questionnaires about socio-demographic characteristics, inclusion and non-inclusion criteria, consent

SECONDARY OUTCOMES:
Description of the patient's hallucinations | 1 day
  Qualitative study of hallucinations (for patients who said they had or had had them during the first interview).
  The Scale used is PSAS : a questionnaire for the characteristics of hallucinations When establishing the protocol, the PSAS (Psycho-Sensory Hallucinations Scale) was chosen because it is one of the only scales studying the different types of hallucinations (auditory, visual, coenesthetic, olfactory and tasteful) validated in French.
Search for dissociative elements | 1 day
  Search for dissociative elements in the patient with the scale: DES-II DES-II is a self-questionnaire to detect individuals with a dissociative disorder or disorder with a high dissociative component, as well as to quantify dissociative experiences. It consists of 28 questions on situations in which the subject indicates, in percentage, the frequency with which each situation occurs.
Investigation of traumatic elements | 1 day
  Investigation of traumatic elements and post-traumatic stress disorder (PTSD) with the scales used: THQ THQ is a self-administered questionnaire consisting of 24 closed questions (yes / no) evaluating the presence of a number of potentially traumatic events in the life of an individual. They are divided into 3 categories (crime, natural disasters and traumas, physical and sexual experiences)
Investigation of traumatic elements | 1 day
  Investigation of traumatic elements and post-traumatic stress disorder (PTSD) with the scales used: PCL-S PCL-S is a self-administered questionnaire that evaluates the symptoms of PTSD. It is translated into French and validated for the detection and monitoring of PTSD. It assesses the existence of PTSD symptoms related to a specific and identified traumatic event. In this study we define the specific traumatic event with the patient before the handover. The questionnaire consists of 17 questions around the main symptoms described by the DSM-IV

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Mathur, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No